CLINICAL TRIAL: NCT03092284
Title: Allogeneic Adipose Tissue-derived Stromal/Stem Cell Therapy in Patients With Ischemic Heart Disease and Heart Failure: A Phase II Danish Multicentre Study
Brief Title: Allogeneic Stem Cell Therapy in Heart Failure
Acronym: CSCC_ASCII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: JKastrup (Other)
Responsible Party: Sponsor-Investigator, JKastrup, Professor Chief Physician, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSCC_ASCII
Record Dates: First submitted 2015-07-20; First posted 2017-03-27 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cardiology Stem Cell Centre Adipose Stem Cell (CSCC_ASC) (Active Comparator): Allogeneic adipose derived stromal cells
  Interventions: Biological: Cardiology Stem Cell Centre Adipose Stem Cell (CSCC_ASC)
- Placebo (Placebo Comparator): Saline
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Cardiology Stem Cell Centre Adipose Stem Cell (CSCC_ASC) — Direct intramyocardial injection of CSCC_ASC
  Arms: Cardiology Stem Cell Centre Adipose Stem Cell (CSCC_ASC)
Biological: Placebo — Saline
  Arms: Placebo

SUMMARY:
The present aim is to perform at clinical double-blind placebo-controlled Cardiology Stem Cell Centre - Adipose Stem Cells (CSCC_ASC) study in heart failure patients to investigate the regenerative capacity of the CSCC_ASC treatment.

DETAILED DESCRIPTION:
The primary objective is to investigate the regenerative capacity of direct intra-myocardial injection of 100 mio. allogeneic CSCC_ASCs in patients with reduced left ventricular Ejection Fraction (EF) (≤45%) and heart failure in a double-blind placebo-controlled design.

A total of 81 patients with will be enrolled in the study and treated in a 2:1 randomization with either CSCC_ASC or placebo (saline).

The primary endpoint is change in left ventricle end-systolic volume (LVESV) at 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. 30 to 80 years of age
2. Signed informed consent
3. Chronic stable ischemic heart disease
4. Symptomatic heart failure - New York Heart Association (NYHA) class II-III
5. EF ≤45%
6. Plasma NT-pro-BNP > 300 pg/ml (> 35 pmol/L) in sinus rhythm and plasma NT-pro-BNP > 422 pg/ml (> 450 pmol/L) in patients with atrial fibrillation
7. Maximal tolerable heart failure medication
8. Medication unchanged two months prior to inclusion
9. No option for percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG)
10. Patients who have had PCI or CABG within six months of inclusion must have a new angiography less than one month before inclusion or at least four months after the intervention to rule out early restenosis
11. Patients cannot be included until three months after implantation of a cardiac resynchronisation therapy device

Exclusion Criteria:

1. Heart Failure (NYHA I or IV)
2. Acute coronary syndrome with elevation of creatine kinase (CK) isoenzyme MB (CKMB) or troponins, stroke or transitory cerebral ischemia within six weeks of inclusion
3. Other revascularisation treatment within four months of treatment
4. If clinically indicated the patient should have a coronary angiography before inclusion
5. Moderate to severe aortic stenosis (valve area < 1.3 mm2) or valvular disease with option for surgery.
6. Diminished functional capacity for other reasons such as: obstructive pulmonary disease (COPD) with forced expiratory volume (FEV) <1 L/min, moderate to severe claudication or morbid obesity
7. Clinical significant anaemia (haemoglobin < 6 mmol/L), leukopenia (leucocytes < 2 109/L), leucocytosis (leucocytes >14 109/L) or thrombocytopenia (thrombocytes < 50 109/L)
8. Anticoagulation treatment that cannot be paused during cell injections
9. Patients with reduced immune response
10. History with malignant disease within five years of inclusion or suspected malignity - except treated skin cancer other than melanoma
11. Pregnant women
12. Other experimental treatment within four weeks of baseline tests
13. Participation in another intervention trial

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2021-07 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
change in left ventricle end-systolic volume (LVESV) from base line to 6 months follow-up measured by echocardiography and computerized tomography | 6 months
  change in left ventricle end-systolic volume (LVESV) from base line to 6 months follow-up measured by echocardiography and computerized tomography

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 12 months
  Safety is evaluated by the incidence and severity of serious adverse events and suspected unrelated serious adverse events at 12 months follow-up
Efficacy left ventricle | 6 months
  change in left ventricle ejection fraction (EF) measured by echocardiography and computerized tomography
Efficacy clinical function assessed by change in Kansas City Cardiomyopathy Questionnaire (KCCQ) from baseline to 6 months follow-up | 6 months
  change in Kansas City Cardiomyopathy Questionnaire (KCCQ) from baseline to 6 months follow-up
Efficacy clinical function assessed by change in Seattle Angina Questionnaire and 6 min walking test from baseline to 6 months follow-up | 6 months
  change in Seattle Angina Questionnaire and 6 min walking test from baseline to 6 months follow-up
Efficacy clinical function assessed by change in 6 min walking test from baseline to 6 months follow-up | 6 months
  change in 6 min walking test from baseline to 6 months follow-up
Efficacy clinical function assessed by change in Kansas City Cardiomyopathy Questionnaire (KCCQ) from baseline to 12 months follow-up | 12 months
  change in Kansas City Cardiomyopathy Questionnaire (KCCQ) from baseline to 12 months follow-up
Efficacy clinical function assessed by change in Seattle Angina Questionnaire and 6 min walking test from baseline to 12 months follow-up | 12 months
  change in Seattle Angina Questionnaire and 6 min walking test from baseline to 12 months follow-up
Efficacy clinical function assessed by change in 6 min walking test from baseline to 12 months follow-up | 12 months
  change in 6 min walking test from baseline to 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kastrup, Professor MD, Study Director — Rigshospitalet, Denmark
Locations (1):
- Cardiac Catheterization Laboratory 2014, The Heart Centre, University Hospital, Rigshospitalet, Copenhagen Ø, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data can be share for scientific collaboration

REFERENCES:
- [Derived] Qayyum AA, Mouridsen M, Nilsson B, Gustafsson I, Schou M, Nielsen OW, Hove JD, Mathiasen AB, Jorgensen E, Helqvist S, Joshi FR, Johansen EM, Follin B, Juhl M, Hojgaard LD, Haack-Sorensen M, Ekblond A, Kastrup J. Danish phase II trial using adipose tissue derived mesenchymal stromal cells for patients with ischaemic heart failure. ESC Heart Fail. 2023 Apr;10(2):1170-1183. doi: 10.1002/ehf2.14281. Epub 2023 Jan 13. PMID 36638837